CLINICAL TRIAL: NCT04467736
Title: A Randomized Controlled Trial Evaluating Hyaluronic Acid As a Wound Healing Agent Following Alveolar Ridge Preservation
Brief Title: Wound Healing with Hyaluronic Acid After Alveolar Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-07718
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healing Wound
Keywords: Alveolar ridge preservation; Hyaluronic acid; Wound healing

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Patients will be randomly allocated to the 'test group (Hyaluronic acid)' or the 'control group (No hyaluronic acid). An equal number of sealed envelopes will be prepared internally labelled as 'test group' or 'control group'. Just after alveolar ridge preservation, a sealed envelope will be randomly selected and opened to reveal further treatment.
  The measuring investigator will not be involved in the treatment of any of the patients and will be blinded to allow unbiased registrations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): No further treatment after alveolar ridge preservation
- Test (Active Comparator): In case the test group comes out, instructions for the daily application of hyaluronic acid (Gengigel Forte©) will be given. Hyaluronic acid will be administered by the patient 3 times per day during 7 days.
  Interventions: Device: Gengigel Forte©

INTERVENTIONS:
Device: Gengigel Forte© — Gengigel (hyaluronic acid) will be administered by the patient 3 times per day during 7 days following alveolar ridge preservation
  Arms: Test

SUMMARY:
After tooth extraction, shrinkage of the bone is expected after 6 months. These changes may hamper dental implant placement and compromise soft tissue aesthetics. Alveolar Ridge Preservation (ARP) includes application of bovine-derived deproteinized bone particles in the extraction site. This technique is widely performed and drastically limits aforementioned volumetric changes.

The amount of bone preservation following ARP is affected by the soft tissue barrier. In an open healing situation, it takes about 4 weeks to have complete soft tissue closure. Faster soft tissue closure could optimize the amount of bone preservation with obvious benefits for implant placement and aesthetics.

Recent presentations showed the application of hyaluronic acid after ARP. However, no evidence can be found in the literature. This study aims to evaluate the wound healing potential of hyaluronic acid following ARP, as this has never been performed, yet seems promising from a biological point of view.

DETAILED DESCRIPTION:
Aim:

This study aims to evaluate the wound healing potential of hyaluronic acid (HA) following alveolar ridge preservation (ARP), as this has never been performed, yet seems promising from a biological point of view.

Sample size calculation:

A sample size calculation using a two-sample pooled t-test was performed in SAS Power and Sample Size based on a comparison of mean overall wound reduction from baseline to 21 days between the control and test group. The calculation was based on finding a mean difference of 20% between these groups with a standard deviation of 21.6 for the control and 21.6 for the test group. A pilot study was executed to obtain these findings as no other data are available. With alpha set at 0.05 and a power of 0.08, the sample size calculation indicated 19 patients to be included per group. To compensate for drop-outs, 25 would be treated with hyaluronic acid and 25 would be treated without.

Clinicians and centers, randomization, allocation concealment and blinding:

3 clinicians linked to the Department of Periodontology and Oral Implantology at UGent - UZ Gent will treat a total of 50 patients. Each clinician will treat at least 10 patients. Patients will be randomly allocated to the 'test group (Hyaluronic acid)' or the 'control group (No hyaluronic acid). An equal number of sealed envelopes will be prepared internally labelled as 'test group' or 'control group'. Just after ARP, a sealed envelope will be randomly selected and opened to reveal further treatment. In case the test group comes out, instructions for the daily application of HA (Gengigel Forte©) will be given. HA will be administered by the patient 3 times per day during 7 days.

The measuring investigator will not be involved in the treatment of any of the patients and will be blinded to allow unbiased registrations.

Surgical procedure:

After screening and having obtained informed consent by the patient, the tooth is extracted and ARP is performed by placing collagen-enriched deproteinized bovine bone mineral (DBBM, Bio-Oss collagen 100 mg or 250 mg, Geistlich Biomaterials, Switserland) in the alveolar socket. Subsequently, a collagen matrix (Mucograft seal, Geistlich Biomaterials, Switserland), is sutured on top to protect the underlying DBBM. At the end of the surgical procedure, the sealed envelope is opened to reveal the allocated treatment and instructions to the patients are given (application of Gengigel Forte© 3 times per day during 7 days).

Intra-surgical registrations:

Intra-surgically, the dimensions of the buccal bone plate will be registered. Papillae are analyzed if they were detached from the bone mesial and distal during extraction. Subsequently, the size of the Mucograft seal (Geistlich Biomaterials, Switserland) is measured. Immediately after ARP, a conebeam computed tomography (CBCT) of the alveolar bone is taken and an intra-oral scan of the soft tissues is performed (for study purposes). Afterwards, an occlusal clinical photograph is taken. The wound dimension is registered by measuring the maximum mesio-distal and bucco-oral dimension of the wound with a periodontal probe to the nearest 0.5 mm (for study purposes).

One-week post-surgery:

One week after ARP, patient's compliance concerning the application of HA 3 times a day is evaluated, as well as the number of painkillers taken. A Visual Analog Scale (VAS) will be filled out by patients to register pain, swelling and bleeding after surgery. (for study purposes) Furthermore, a socket wound healing scoring (SWHS, is given to each extraction wound and another occlusal photograph is taken at the end of the consultation. To evaluate the soft tissue closure, the maximum mesio-distal and bucco-oral dimension of the remaining wound is measured with a periodontal probe to the nearest 0.5 mm. (for study purposes)

Wound closure after 21 days:

Three weeks post-surgery, the maximum mesio-distal and bucco-oral dimension of the remaining wound is measured with a periodontal probe to the nearest 0.5 mm. For each aspect (mesio-distal and bucco-oral) the percentage wound reduction is calculated as follows:

100 - ((Maximum wound dimension after 21 days * 100) / maximum wound dimension immediately after ARP)

The overall wound reduction is calculated as follows:

(Wound reduction at the mesio-distal aspect + wound reduction at the bucco-oral aspect) / 2

SWHS is determined for each wound. Finally, an occlusal clinical photograph is taken.

4 months after surgery: An occlusal photograph is taken to analyze mucosal scarring using the Mucosal Scarring Index (MSI, for study purposes). A second CBCT is made to measure dimensional changes of the alveolar process. A second intra-oral scan is made to measure dimensional changes in buccal soft tissue profile. (standard of care)

Data analysis:

Depending on the distribution of the data, an independent samples t-test or Mann-Whitney U test will be performed on the following parameters:

* Wound reduction after 21 days (primary outcome)
* VAS swelling
* VAS pain
* Number of painkillers consumed
* Socket Wound healing score
* Mucosal scarring index
* Dimensional changes in the buccal soft tissue profile
* Dimensional changes of the alveolar process

For the following categorical variables, a Fisher's exact will be performed:

* Compliance
* Bleeding

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Good oral hygiene defined as a full-mouth plaque score ≤25%;
* One or two neighboring teeth;
* Need for ARP after tooth extraction with >50% buccal bone still present

Exclusion Criteria:

* Systemic diseases;
* Smoking;
* (History) of periodontal disease;
* Untreated caries lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Wound reduction | Week 3 after ARP
  performed by measuring the maximum mesio-distal and bucco-oral dimension of the wound immediately after ARP and after 21 days

SECONDARY OUTCOMES:
Compliance | Week 1
  patients will be asked if they applied HA 3 times a day as prescribed? Protocol violations will be recorded to see if they have an impact on the outcome (fully compliant patients versus weakly compliant patients).
Number of painkillers consumed | Week 1
VAS pain | Week 1
  Visual Analogue Scale for pain: the patient has to indicate the intensity of pain perception during the first week after surgery on a 10 cm line
VAS swelling | Week 1
  Visual Analogue Scale for swelling: the patient has to indicate the amount of swelling perception during the first week after surgery on a 10 cm line
Bleeding | Week 1
  Patients will be asked if they experienced post-operative bleeding
Socket wound healing score | Week 1 and 3
  This index will be used to assess wound dehiscence, epithelialization, quality of granulation tissue filling the post-extraction socket, and depth between early granulation tissue and wound margin.
  Assessments will be performed at performed at 7 and 21 days following surgery using a blunt periodontal probe with millimetric markers and scored as a number between 0 (best) and 4 (worst). In contrast to the study from (Afat et al., 2018), this study will not probe inside the healing wound.
Mucosal scarring index | 4 months
  The MSI is a composite index based on five parameters: width, height/contour, color, suture marks, and overall appearance. Each parameter is assessed with a 0-1-2 score, yielding an MSI score ranging from 0 (no scar) to 10 (most extreme scar)
Dimensional changes in the buccal soft tissue profile | At time of surgery and at 4 months
  Immediately after surgery and at 4 months an intra-oral optical scan of the implant site and neighboring teeth will be taken (Trios, 3shape, Copenhagen, Denmark). The region of interest (ROI) will be defined on the 4-month STL files with a trapezoid shape encompassing the following borders (fig. 2): 0.5 mm apical to the midfacial soft tissue level (coronal), 4 mm apical and parallel to the first line (apical), mesial and distal line angle. This ROI may vary between patients due to anatomical variation but will be kept constant in each patient and site over time. The STL images of baseline and follow-up will be superimposed and matched using the best-fit algorithm at the adjacent tooth surfaces. The linear changes in BSP will be calculated by the software and expressed in mm corresponding to the mean distance between the surfaces representing the evaluated time points.
Dimensional changes of the alveolar process | Immediately after surgery and at 4 months
  Comparing CBCT-scan after surgery and after 4 months. First, a line parallel and perpendicular to the tooth axis is drawn. Hereby, bone dimensions can be measured at different vertical heights on the alveolar process. The level of the palatal bone crest at T0 is used as a reference line (level 0). The horizontal dimension of the process is registered at 1, 3, and 5 mm apical to the reference line (level -1, -3, and -5). After performing all measurements on the baseline CBCT (T0), the software will be switched to the superimposed image (T1) so that the measurements can be performed while using the same reference levels

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afat IM, Akdogan ET, Gonul O. Effects of Leukocyte- and Platelet-Rich Fibrin Alone and Combined With Hyaluronic Acid on Pain, Edema, and Trismus After Surgical Extraction of Impacted Mandibular Third Molars. J Oral Maxillofac Surg. 2018 May;76(5):926-932. doi: 10.1016/j.joms.2017.12.005. Epub 2017 Dec 13. PMID 29304325
- [Background] Afat IM, Akdogan ET, Gonul O. Effects of leukocyte- and platelet-rich fibrin alone and combined with hyaluronic acid on early soft tissue healing after surgical extraction of impacted mandibular third molars: A prospective clinical study. J Craniomaxillofac Surg. 2019 Feb;47(2):280-286. doi: 10.1016/j.jcms.2018.11.023. Epub 2018 Dec 3. PMID 30579747
- [Background] Cosyn J, Cleymaet R, De Bruyn H. Predictors of Alveolar Process Remodeling Following Ridge Preservation in High-Risk Patients. Clin Implant Dent Relat Res. 2016 Apr;18(2):226-33. doi: 10.1111/cid.12249. Epub 2014 Jul 17. PMID 25041378
- [Background] Eskandarinia A, Kefayat A, Gharakhloo M, Agheb M, Khodabakhshi D, Khorshidi M, Sheikhmoradi V, Rafienia M, Salehi H. A propolis enriched polyurethane-hyaluronic acid nanofibrous wound dressing with remarkable antibacterial and wound healing activities. Int J Biol Macromol. 2020 Apr 15;149:467-476. doi: 10.1016/j.ijbiomac.2020.01.255. Epub 2020 Jan 27. PMID 32001284
- [Background] Hammerle CH, Araujo MG, Simion M; Osteology Consensus Group 2011. Evidence-based knowledge on the biology and treatment of extraction sockets. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:80-2. doi: 10.1111/j.1600-0501.2011.02370.x. PMID 22211307
- [Background] Litwiniuk M, Krejner A, Speyrer MS, Gauto AR, Grzela T. Hyaluronic Acid in Inflammation and Tissue Regeneration. Wounds. 2016 Mar;28(3):78-88. PMID 26978861
- [Background] Neuman MG, Nanau RM, Oruna-Sanchez L, Coto G. Hyaluronic acid and wound healing. J Pharm Pharm Sci. 2015;18(1):53-60. doi: 10.18433/j3k89d. PMID 25877441
- [Background] Seyssens L, Eghbali A, Christiaens V, De Bruyckere T, Doornewaard R, Cosyn J. A one-year prospective study on alveolar ridge preservation using collagen-enriched deproteinized bovine bone mineral and saddle connective tissue graft: A cone beam computed tomography analysis. Clin Implant Dent Relat Res. 2019 Oct;21(5):853-861. doi: 10.1111/cid.12843. Epub 2019 Aug 28. PMID 31456345
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Background] Wessels R, De Roose S, De Bruyckere T, Eghbali A, Jacquet W, De Rouck T, Cosyn J. The Mucosal Scarring Index: reliability of a new composite index for assessing scarring following oral surgery. Clin Oral Investig. 2019 Mar;23(3):1209-1215. doi: 10.1007/s00784-018-2535-6. Epub 2018 Jul 3. PMID 29971512
- [Background] Yildirim S, Ozener HO, Dogan B, Kuru B. Effect of topically applied hyaluronic acid on pain and palatal epithelial wound healing: An examiner-masked, randomized, controlled clinical trial. J Periodontol. 2018 Jan;89(1):36-45. doi: 10.1902/jop.2017.170105. PMID 28914592
- [Background] Zeltner M, Jung RE, Hammerle CH, Husler J, Thoma DS. Randomized controlled clinical study comparing a volume-stable collagen matrix to autogenous connective tissue grafts for soft tissue augmentation at implant sites: linear volumetric soft tissue changes up to 3 months. J Clin Periodontol. 2017 Apr;44(4):446-453. doi: 10.1111/jcpe.12697. Epub 2017 Feb 11. PMID 28107560
- [Derived] Eeckhout C, Ackerman J, Glibert M, Cosyn J. A randomized controlled trial evaluating hyaluronic acid gel as wound healing agent in alveolar ridge preservation. J Clin Periodontol. 2022 Mar;49(3):280-291. doi: 10.1111/jcpe.13589. Epub 2021 Dec 30. PMID 34961942